CLINICAL TRIAL: NCT02986867
Title: SAbR-Induced Innate Immunity in Urothelial Carcinoma, Melanoma, and Cervical Carcinoma
Brief Title: SAbR Induced Innate Immunity in Urothelial Carcinoma, Melanoma, and Cervical Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU 092016-055
Record Dates: First submitted 2016-11-21; First posted 2016-12-08 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Urothelial Carcinoma; Melanoma; Cervical Carcinoma in Situ
MeSH Terms: conditions — Carcinoma, Transitional Cell; Melanoma; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SAbR (Experimental): SAbR treatment of lesions
  Interventions: Radiation: SAbR Treatment of Lesions

INTERVENTIONS:
Radiation: SAbR Treatment of Lesions — SAbR will be administered as per the guidelines of UTSW with a single 24-27Gy or three 10-14 Gy/fraction fractions totaling 33-48Gy. Lesions receiving SAbR will be called "radiated" lesions.

SUMMARY:
The study is an exploratory prospective, single center study with correlative endpoints. The study will investigate the association of tumor cGAS STING signaling with SAbR. Tumor core biopsies will be processed and analyzed as described above. Medical records electronic medical records will be used to collect demographic and medical information and imaging studies.

DETAILED DESCRIPTION:
Within 2 weeks of planned SAbR, patients will have a core biopsy of the lesion to receive SAbR. Laboratory values will be obtained prior to biopsy. Once the laboratory values are found to be within the safe margin for biopsy, multiple (approximately 5) core biopsies will be obtained with an 18-guage or 19-gauge needle under CT or US guidance. Tissue will be snap frozen with liquid nitrogen and immediately transferred to the laboratory of Dr. Zhijian "James" Chen, PhD, Professor, Department of Molecular Biology.

SAbR will be administered as per the guidelines of UTSW with a single 24-27Gy or three 10-14 Gy/fraction fractions totaling 33-48Gy. Lesions receiving SAbR will be called "radiated" lesions. Prior irradiated lesions will be excluded. SABR will be administered within 2 weeks of the study initial core biopsy. The SAbR dose and fractionation scheme is generated to deliver a potent dose to ablate the targeted lesions and at the same time maximize an immune response. Since multiple studies have shown an influx of lymphocytes and monocytes after tumor irradiation and since these cells play a critical role in antigen presentation and initiation of an adaptive immune response, multiple fraction irradiation which would kill these infiltrating immunocytes, is discouraged. Therefore a single fraction or a three fraction treatment regimen is recommended, and a single fraction treatment is preferred over three fractions. Due to normal organ toxicity and limits of dose constraints, sometimes a three fraction treatment must be undertaken and in those cases it is recommended that the treatment course is completed within 7-10 days-preferably 5 business days. Radiation dose-immune response studies have shown a linear increase in immune response with increased dose per fraction of radiation without demonstration of a plateau. Two studies comparing 15Gy x 1 vs 5Gy x3, and 20Gy x1 vs 5Gy x4 have shown a superior immune response generated by the single fraction radiation. Clinical experience with oligometastatic patients treated at 1-5 sites of disease has also showed an increase in progression-free survival with the increasing radiation dose per fraction. A dose of less than 7.5 Gy per fraction has demonstrated lower induction of systemic IFN-γ producing cells, and a previous phase II study of mRCC patients treated with HD IL-2 and singe fraction of 8Gy irradiation to a single lesion did not show an overall improvement in response rate. Therefore 8Gy per fraction is the lowest permitted dose for this study and can be used only when administering the three fraction regimen as described in the prescription dose table below. Investigators will have discretion in choosing from either of the biologically equivalent dose levels using one or three fractions, although a single fraction is preferred over three fraction treatments. Treating physician will have further discretion in selecting the number and location of sites to treat if multiple sites of disease are present. Maximum number of lesions treated is deemed as feasible per the treating radiation oncologist. However, for the purposes of this protocol, only a single site will be studied and must be safely amenable to repeat core biopsy. Thus, the single site for the study will be either in subcutaneous tissues, nodes, isolated masses or liver. The gross target/tumor volume--GTV should be at least 2 cm3 in size, corresponding to roughly a 1.5 cm diameter tumor. This is to ensure that adequate tumor volume for therapy and for biopsy and therefore adequate tumor cells roughly 108 -109 cells/cm3 are killed for antigen presentation. Treating physicians should choose their dose based on established planning guidelines at their center including their ability to respect normal tissue tolerance.

Within 24 + 6 hours of the first SAbR, a second core biopsy of the "target" irradiated lesion will be performed identically to the first biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of advanced/metastatic urothelial carcinoma, melanoma, or cervical carcinoma.
* Planned treated with SAbR.
* Age greater than or equal to 18 years.
* Lesion to receive SAbR safely accessible for core biopsy-mass >1.5cm diameter and located in node, liver, or soft tissues.
* Hgb >10g/dL before or after transfusion.
* Platelets >50,000/L
* INR <1.5
* If contrast enhanced CT needed to locate the lesion for core biopsy, then derived creatinine clearance >30cc/min
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior radiation therapy to target lesion.
* Target lesion not safely accessible for core biopsies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Comparison of immune checkpoint treated tumors | 36 months
  Compare cGAMP levels, interferon response gene expression and phospho-STING in tumors of immune checkpoint treated patients.
SAbR effects on cGAMP in tumors | 36 months
  Number of participants with SAbRrelated tumor changes indicated by cGAMP in comparison to Baseline.
SAbR effects on interferon response in tumors | 36 months
  Number of participants with SAbRrelated tumor changes indicated by interferon response mRNAs in comparison to Baseline.
SAbR effects on phosphor-STING in tumors | 36 months
  Number of participants with SAbRrelated tumor changes indicated by phospho-STING in comparison to Baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No